CLINICAL TRIAL: NCT06463717
Title: Comparing the Efficacy and Safety of Autologous Hematopoietic Stem-cell Transplantation Versus Non Transplantation Regimen in Primary Multiple Myeloma Achieved MRD Negativity After Induction: A Multiple Center, Prospective Cohort Study
Brief Title: Primary Multiple Myeloma Who Achieved MRD Negativity After Induction Therapy, ASCT or Not
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other); The Affiliated Hospital of Medical College, Ningbo University (Other); Dongyang People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IIT20230339B-R1
Record Dates: First submitted 2024-06-05; First posted 2024-06-18 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2023-12

CONDITIONS: Multiple Myeloma; Minimal Residual Disease
Keywords: Minimal Residual Disease Negativity; Autologous Stem Cell Transplantation
MeSH Terms: conditions — Multiple Myeloma; Neoplasm, Residual | interventions — Transplantation, Autologous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASCT regimen: Primary multiple myeloma patients who receive autologous hematopoietic stem-cell transplantation (ASCT) after they achieved MRD negativity after induction
  Interventions: Drug: Transplant, Autologous
- non ASCT regimen: Primary multiple myeloma patients who receive non autologous hematopoietic stem-cell transplantation (ASCT) regimen such as 4-6 cycles of bortezomib-lenalidomide-dexamethasone after they achieved MRD negativity after induction
  Interventions: Drug: Chemotherapy drug

INTERVENTIONS:
Drug: Transplant, Autologous — High-dose melphalan followed by autologous stem cell transplantation
  Other Names: ASCT
  Groups: ASCT regimen
Drug: Chemotherapy drug — Regimen such as Bortezomib plus Lenalidomide plus Dexamethasone
  Other Names: Non ASCT regimen
  Groups: non ASCT regimen

SUMMARY:
The goal of this observational study is to compare the efficacy and safety of autologous hematopoietic stem-cell transplantation (ASCT) versus non ASCT regimens in primary multiple myeloma patients achieved MRD negativity after induction.

The main question it aims to answer is:

In primary multiple myeloma patients who achieved MRD negativity after induction, non ASCT regimens are not inferior to ASCT or not? Participants will receive ASCT or non ASCT regimen according to their own choice.

Researchers will compare ASCT and non ASCT group see if any significant difference in efficacy and safety.

DETAILED DESCRIPTION:
Background Multiple myeloma (MM) is third most common hematological malignancy. For newly diagnosed MM patients who are transplantation eligible, the current standard treatment regimen is induction therapy with bortezomib plus lenalidomide plus dexamethasone (VRD), high-dose melphalan (200 mg/m2) followed by autologous stem cell transplantation (MEL200-ASCT), and maintenance therapy with lenalidomide and/or proteasome inhibitors. However, MEL200-ASCT requires hospitalization and may induces toxic side effects. In recent years, multiple MM international research centers have explored and compared the efficacy of different treatment regimens (such as bortezomib plus melphalan plus prednisone, bortezomib plus lenalidomide plus dexamethasone, carfilzomib plus cyclophosphamide plus dexamethasone, and carfilzomib plus lenalidomide plus dexamethasone) with MEL200-ASCT, and found that MEL200-ASCT has a higher progression free survival compared to the aforementioned chemotherapy regimens, but failed to show benefit in overall survival. The advantage of MEL200-ACT in progression free survival can be attributed to its ability to achieve deeper therapeutic responses compared to chemotherapy regimens, including a higher complete response (CR), very good partial response (VGPR), and a higher negative rate for minimal residual disease (MRD) or sustained negative rate for MRD.

MRD was introduced by the International Myeloma Working Group in 2016, which implies deeper clinical response than CR and can be detected by flow cytometry or second-generation sequencing, with a sensitivity of at least 10-5. Research has shown that MRD is the most powerful prognostic factor for MM, and MM patients with negative MRD have a significant superior survival than MRD positive patients. As mentioned earlier, MEL200-ASCT induces deeper therapeutic response than chemotherapy, and results in superior progression survival. So, in patients who have already reached MRD negative after VRD induction treatment, does MEL200-ASCT still have an advantage in progression free survival compared to chemotherapy? A study comparing the efficacy of MEL200-ASCT with carfilzomib plus cyclophosphamide and dexamethasone found that among patients with detectable MRD after induction therapy, MEL200-ASCT group had a higher progression free survival rate than chemotherapy. However, there was no evidence suggesting that MEL200-ASCT is beneficial for patients who have already obtained MRD negative after induction therapy.

Therefore, this study aims to investigate the status of MEL200-ACT in newly diagnosed MM patients who have achieved MRD negative after induction therapy with the current standard protocol.

Data collection Patient who met the enrollment criteria is unselected recorded and followed regularly.

Sample size calculation This study aims to demonstrate that non ASCT regimens is not inferior to high dose melphalan followed by ASCT in terms of progression free survival in MM patients who already obtained MRD negative after induction therapy. Based on available date, 2-year progression free survival rate was 85% for patients received MRD negativity after induction therapy and followed by ASCT. Therefore, the investigators assure that 2-year progression free survival rate of non ASCT regimen group should not be less than 75%, i.e. a non-inferiority margin of 10%. Using a one-sided non-inferiority test for two exponential survival curves with 0.025 alpha, 0.8 power, a common exponential dropout rate of 10% and number of non ASCT and ASCT patients in a 3:2 ratio, 126 patients for non ASCT and 84 patients for ASCT group are required.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed multiple myeloma according to the criteria of International Working Group of Myeloma
2. Age ranges from 18-70 years old
3. Achieved MRD negativity and at least very good partial response in clinical response after 4-6 courses of induction therapy. MRD is measured by MRD by multicolor flow with a sensitivity of 10-5.
4. At enrollment, score of Eastern Cooperative Oncology Group (ECOG) should be 0-2.
5. Organ function requirement: Blood bilirubin ≤ 2mg/dL (35 μ mol/L), Alanine aminotransferase/Aspartate aminotransferase below 2 times the upper limit of normal value, Creatinine clearance rate (Ccr) ≥ 30ml/min and Cardiac ejection fraction ≥50%.
6. Expected survival more than 3 months.

Exclusion Criteria:

1. Two or more high-risk cytogenetic abnormalities, including del (17p), t (4; 14), t (14; 16), del (1p), amp (1q). Fluorescence in situ hybridization was used to analyze CD138 positive sorted cells, with cut off value of 15% for translocation, 10% for deletion, and amp (1q) of 20%.
2. Extracellular plasma cell disease, central invasion of myeloma, plasma cell leukemia
3. History of other malignant tumors within the past 5 years
4. Patients with HIV, active tuberculosis, clinically active hepatitis A, B, or C
5. Other serious condition that may restrict patients from continuing treatment (such as advanced infection, uncontrolled diabetes, severe cardiac insufficiency, or angina pectoris)
6. General condition not suitable for chemotherapy
7. Pregnant or lactating women
8. Suffering from other serious organic diseases and mental disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary multiple myeloma who achieved MRD negativity after induction therapy are screened by the eligibility Criteria
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 2-year
  Progression-free survival is defined as the duration from diagnosis to the date of death, initial progression, or the last follow-up

SECONDARY OUTCOMES:
sustain MRD negativity | 1-year, 2-year
  The proportion of patients who are still MRD negative at 1-year, 2-years after achieving MRD negativity after induction therapy
Number of Participants With Treatment-Related Adverse Events | Once enrolled, an average of 2 year
  All adverse events and second primary malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Meng, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gay F, Musto P, Rota-Scalabrini D, Bertamini L, Belotti A, Galli M, Offidani M, Zamagni E, Ledda A, Grasso M, Ballanti S, Spadano A, Cea M, Patriarca F, D'Agostino M, Capra A, Giuliani N, de Fabritiis P, Aquino S, Palmas A, Gamberi B, Zambello R, Petrucci MT, Corradini P, Cavo M, Boccadoro M. Carfilzomib with cyclophosphamide and dexamethasone or lenalidomide and dexamethasone plus autologous transplantation or carfilzomib plus lenalidomide and dexamethasone, followed by maintenance with carfilzomib plus lenalidomide or lenalidomide alone for patients with newly diagnosed multiple myeloma (FORTE): a randomised, open-label, phase 2 trial. Lancet Oncol. 2021 Dec;22(12):1705-1720. doi: 10.1016/S1470-2045(21)00535-0. Epub 2021 Nov 11. PMID 34774221
- [Background] Cavo M, Gay F, Beksac M, Pantani L, Petrucci MT, Dimopoulos MA, Dozza L, van der Holt B, Zweegman S, Oliva S, van der Velden VHJ, Zamagni E, Palumbo GA, Patriarca F, Montefusco V, Galli M, Maisnar V, Gamberi B, Hansson M, Belotti A, Pour L, Ypma P, Grasso M, Croockewit A, Ballanti S, Offidani M, Vincelli ID, Zambello R, Liberati AM, Andersen NF, Broijl A, Troia R, Pascarella A, Benevolo G, Levin MD, Bos G, Ludwig H, Aquino S, Morelli AM, Wu KL, Boersma R, Hajek R, Durian M, von dem Borne PA, Caravita di Toritto T, Zander T, Driessen C, Specchia G, Waage A, Gimsing P, Mellqvist UH, van Marwijk Kooy M, Minnema M, Mandigers C, Cafro AM, Palmas A, Carvalho S, Spencer A, Boccadoro M, Sonneveld P. Autologous haematopoietic stem-cell transplantation versus bortezomib-melphalan-prednisone, with or without bortezomib-lenalidomide-dexamethasone consolidation therapy, and lenalidomide maintenance for newly diagnosed multiple myeloma (EMN02/HO95): a multicentre, randomised, open-label, phase 3 study. Lancet Haematol. 2020 Jun;7(6):e456-e468. doi: 10.1016/S2352-3026(20)30099-5. Epub 2020 Apr 30. PMID 32359506
- [Background] Attal M, Lauwers-Cances V, Hulin C, Leleu X, Caillot D, Escoffre M, Arnulf B, Macro M, Belhadj K, Garderet L, Roussel M, Payen C, Mathiot C, Fermand JP, Meuleman N, Rollet S, Maglio ME, Zeytoonjian AA, Weller EA, Munshi N, Anderson KC, Richardson PG, Facon T, Avet-Loiseau H, Harousseau JL, Moreau P; IFM 2009 Study. Lenalidomide, Bortezomib, and Dexamethasone with Transplantation for Myeloma. N Engl J Med. 2017 Apr 6;376(14):1311-1320. doi: 10.1056/NEJMoa1611750. PMID 28379796
- [Background] Yong K, Wilson W, de Tute RM, Camilleri M, Ramasamy K, Streetly M, Sive J, Bygrave CA, Benjamin R, Chapman M, Chavda SJ, Phillips EH, Del Mar Cuadrado M, Pang G, Jenner R, Dadaga T, Kamora S, Cavenagh J, Clifton-Hadley L, Owen RG, Popat R. Upfront autologous haematopoietic stem-cell transplantation versus carfilzomib-cyclophosphamide-dexamethasone consolidation with carfilzomib maintenance in patients with newly diagnosed multiple myeloma in England and Wales (CARDAMON): a randomised, phase 2, non-inferiority trial. Lancet Haematol. 2023 Feb;10(2):e93-e106. doi: 10.1016/S2352-3026(22)00350-7. Epub 2022 Dec 15. PMID 36529145
- [Background] Kumar S, Paiva B, Anderson KC, Durie B, Landgren O, Moreau P, Munshi N, Lonial S, Blade J, Mateos MV, Dimopoulos M, Kastritis E, Boccadoro M, Orlowski R, Goldschmidt H, Spencer A, Hou J, Chng WJ, Usmani SZ, Zamagni E, Shimizu K, Jagannath S, Johnsen HE, Terpos E, Reiman A, Kyle RA, Sonneveld P, Richardson PG, McCarthy P, Ludwig H, Chen W, Cavo M, Harousseau JL, Lentzsch S, Hillengass J, Palumbo A, Orfao A, Rajkumar SV, Miguel JS, Avet-Loiseau H. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. Lancet Oncol. 2016 Aug;17(8):e328-e346. doi: 10.1016/S1470-2045(16)30206-6. PMID 27511158